CLINICAL TRIAL: NCT05573308
Title: Optimizing Clear Aligners Efficiency With Remote Dental Monitoring and Artificial Intelligence Algorithms
Brief Title: Optimizing Orthodontic Appliances Efficiency With Remote Dental Monitoring and Artificial Intelligence Algorithms
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: American Association of Orthodontists Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Protocol # 2021-0644
Record Dates: First submitted 2022-09-21; First posted 2022-10-10 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Malocclusion; Misaligned Teeth
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Clear Aligners with Dental Monitoring (Experimental): Experiment group: DM (Remote Dental Monitoring approach). Remote Dental Monitoring by DMTM will be implemented in the patient's orthodontic treatment. Pretreatment, 3D digital intra-oral scans will be uploaded to the DMTM dashboard, so they serve as the baseline for 3D tracking of tooth movement. Patients will be trained on how to use the DMTM application and do DM remote scans using their smartphones DM scan box and rector.
  They will be instructed to do the DM scan after the initial tray insertion. Replacement of the aligners trays will be based on DM GO tracking function, which is specifically targeted at clear aligner treatment.
  Interventions: Device: Clear Aligners with Dental Monitoring
- Clear Aligners replaced every 7 days (Active Comparator): Group 2:Control group. All subjects will have conventional aligner treatment with aligners replaced every 7 days, and standard in-office visits every 8 weeks.
  Interventions: Device: Clear Aligners
- Clear Aligners replaced every 14 days (Active Comparator): Group 3: (n=40) Control group. All subjects will have conventional aligner treatment with aligners replaced every 14 days, and standard in-office visits every 8 weeks.
  Interventions: Device: Clear Aligners

INTERVENTIONS:
Device: Clear Aligners with Dental Monitoring — Dental Monitoring™ (DM ™). This digital technology software allows orthodontists to monitor patients remotely through continuous analytics using control vision technology, metaheuristics, and artificial intelligence.31 This app utilizes a patented artificial intelligence machine learning algorithm to calculate 3-dimensional (3D) tooth movements from intraoral photos and videos that patients capture using their smartphone cameras.
  Arms: Clear Aligners with Dental Monitoring
Device: Clear Aligners — Removabale orthodontics appliances
  Arms: Clear Aligners replaced every 14 days; Clear Aligners replaced every 7 days

SUMMARY:
The decision on aligner changing is based on orthodontists' personal experience and common knowledge that an approximated time span for the aligner have exhausted its biological efficacy. However, a one size fits all approach is not always ideal, as an average determined time is not taken into account of a patient's individual biological response. The aligners could be progressed earlier than the determined time, or they may stay inactive for a while, waiting for the in-office visit. Dental MonitoringTM is the only available technology that provides 3D monitoring of teeth movement, reconstructs 3D digital models remotely, and auto-detect clinical situations by their patented AI algorithms. The investigators have reported high accuracy of DMTM to monitor the tooth movement in vitro. However, the efficacy of DMTM on orthodontic treatment and the accuracy of DMTM in the orthodontic patients has not been investigated yet. In this proposal, the investigators are implementing the Dental MonitoringTM application and 3D tracking of tooth movement powered by AI algorisms as a novel tool to customize aligner changing intervals. The ultimate goal is to reduce in-office visits and treatment duration while maintaining regular monitoring, thus not jeopardizing expected results. It is imperative to investigate the Teledentistry for its effectiveness, reliability, ease of use, patient satisfaction, and value on the overall health and oral health system, especially as a critical tool during public health emergency situations.

DETAILED DESCRIPTION:
Specific Aims

Clear Aligners:

To evaluate the effects of implementing Remote Dental Monitoring in orthodontic treatment with clear Aligners. The outcome measures are treatment effectiveness, rate of aligner changing, number of refinements (ratio of added Aligners/planned Aligners- need for midcourse correction), number of appointments, Cost-effectiveness, and patient satisfaction.

Hypothesis 1: Remote Dental Monitoring provides a viable option for continuing good quality of care without compromising the treatment outcome and satisfaction. There are no differences in treatment quality, value, effectiveness, and safety between Remote Dental Monitoring and in-office treatment approaches.

Hypothesis 2: Remote Dental Monitoring can guide the rate of aligner replacement and optimize the treatment.

Hypothesis 3: Remote Dental Monitoring can Improve patient compliance and motivate patients' oral hygiene maintenance

ELIGIBILITY:
Inclusion Criteria:

* Patients who request clear aligner treatment with the sole aim of correcting dental alignment.
* Patients must be 12 years old or older.
* Complete permanent dentition (excluding third molars).
* Non-extraction treatment,
* Upper or lower labial segment crowding. malocclusion to be treated with more than 20 Clear Aligners.

Exclusion Criteria:

* Patients with systematic diseases or syndromes
* Patients with a history or current use of Bisphosphonates
* Patients with current use of nonsteroidal anti-inflammatory drugs (NSAIDs)
* Active periodontal disease
* Presence of dental prostheses,
* The presence of dental anomalies (7) The treatment combined with fixed appliances or other auxiliary appliances.

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-10-17 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
The number of aligners trays completed with an adequate fit | 6 to 30 months
  The primary outcome, the number of trays completed with an adequate fit after 6, 12 months and end of treatment (treatment length ranged 18-30) months.
Number of refinements plans | 6 to 30 months
Number of refinement aligners | 6 to 30 months
The ratio of added trays(refinement)/planned trays. | 6 to 30 months

SECONDARY OUTCOMES:
ABO Discrepancy Index | 6 to 30 months
  The higher the ABO DI score, the more complex the case. Therefore with treatment progress, the DI Score should Decrease at least 1 point from the ABO DI score before treatment.
The American Board of Orthodontics (ABO) Objective grading system (OGS) | 6 to 30 months
  The ABO score for the case is calculated by summing the scores for the 8 categories. The casts are scored in 7 categories (alignment, marginal ridges, buccolingual inclinations, occlusal relationships, occlusal contacts, overjet, and interproximal contacts), and panoramic radiographs are scored according to the single category of root angulation.
  If fewer than 20 points are scored overall, the case is considered to meet the ABO standard. If 20 to 29 points are scored, then the standard of work is undetermined. If more than 30 points are scored, the case is considered unacceptable.
Degree of tooth movement | 6 to 30 months
  3D Comparison Analysis will be performed to evaluate the treatment progress using a sophisticated processing software package (Control; Geomagic, Research Triangle Park, NC). Furthermore, each 3D digital dental scan at T3 will be superimposed on the 3D Digital model of the corresponding treatment stage in the aligner software (representing the ideal outcome).To determine the degree of tooth movement achieved with respect to the prescription, the following formula will be applied to each movement of each tooth.
  1-(Ideal outcome-treatment outcome)/(Ideal outcome- Pre-treatment)

OTHER OUTCOMES:
Number of office visits | 6 to 30 months
  Number of office visits needed to finish the treatment
Patient compliance | 6 to 30 months

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Orthodontic Specialists of Lake County (Antioch), Antioch, Illinois
  - Department of Orthodontics, College of Dentistry University of Illinois Chicago, Chicago, Illinois
  - Orthodontic Specialists of Lake County (Grayslake), Grayslake, Illinois
  - Orthodontic Specialists of Lake County (Gurnee), Gurnee, Illinois

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Morris RS, Hoye LN, Elnagar MH, Atsawasuwan P, Galang-Boquiren MT, Caplin J, Viana GC, Obrez A, Kusnoto B. Accuracy of Dental Monitoring 3D digital dental models using photograph and video mode. Am J Orthod Dentofacial Orthop. 2019 Sep;156(3):420-428. doi: 10.1016/j.ajodo.2019.02.014. PMID 31474272